CLINICAL TRIAL: NCT06872541
Title: Evaluation of Platelet Aggregability in Patients with Non-small Cell Lung Carcinomas
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jose Carlos Nicolau, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5788/23/190
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Assessment of Platelet Aggregability in Patients Patients with Non-small Cell Lung Carcinoma
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (group 1) (Active Comparator): patients without NSCLC and matched by age, sex and presence or absence of smoking in the 6 months before inclusion
  Interventions: Drug: Clopidogrel
- case (group 2) (Active Comparator): patients with NSCLC and matched by age, sex and presence or absence of smoking in the 6 months prior to inclusion
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg uma vez ao dia durante 14 dias

SUMMARY:
Cancer patients are at greater risk of experiencing events thrombotic, arterial or venous, during the course of the disease. Specifically in lung cancer, patients are seven times more prone to developing venous thrombosis, when compared to general population. Platelets influence cancer progression and Tumor microenvironment facilitates platelet activation. Therefore, the main objective of this project is to evaluate platelet aggregation analyzed by aggregometry optics with the use of AggRAM® equipment in patients diagnosed recent non-small cell lung carcinomas, prior to any oncological treatment. Among the secondary objectives, it stands out analyze the primary objective using the PPAnalysis® method (method in developed by our group in partnership with the University of Readings (UK), Plateletworks® and Chrono-log. This is a case-control study, with groups differentiated by the presence or absence of malignant lung neoplasia and matched by age, sex and presence or absence of smoking in the previous 6 months to inclusion. Patients diagnosed with non-cell lung carcinoma Small children without prior treatment will be candidates for participation in the study.

It is expected that at the end important aspects related to aggregation platelet disease are better characterized in this neoplasm, the most important cause of death from cancer in the world, and therapeutic strategies to improvement in morbidity and mortality in the disease can be developed.

DETAILED DESCRIPTION:
Cancer patients are at increased risk of thrombotic complications, especially venous thromboembolism (VTE). The oncology population is seven times more likely to develop thrombosis when compared to the general population, with an incidence of up to 20% of patients during follow-up. It is suggested that the reasons for this greater thrombotic risk are immobility, invasive procedures and changes in coagulation, in addition to possible disorders of platelet aggregation and endothelial function.

The literature suggests that the basic thromboembolic mechanism would be related to the production, by tumor cells, of pro-coagulant factors such as tissue factor and neoplastic pro-coagulant. PAI-1, the main inhibitor of the plasminogen activator pathway, is also produced by tumor cells. Still, tumor production of factors inhibiting the fibrinolytic system plays a role in hypercoagulability and may contribute to tumor angiogenesis. Regarding arterial thrombotic events, although there is no unanimity regarding the causal relationship between the pathologies, epidemiological data strongly suggest that this complication is more common in patients with cancer, compared to the population without the disease.

It is worth mentioning that lung cancer is the most common cause of cancer deaths in the world. It is possible that the high mortality from lung cancer is related, at least partially, to the higher incidence of thrombotic complications presented by these patients, compared to those with other types of cancer. Although VTE is one of the main causes of morbidity and mortality in cancer patients, the use of anticoagulants as primary prophylaxis is not routinely recommended.

The pathophysiological mechanisms involved in the increased risk of thromboembolic events in cancer patients, especially with lung cancer, which, as mentioned, present, in addition to the aggressiveness of the disease itself, a higher incidence of thrombotic events, are still little known. The main objective of this project is to contribute to a better understanding of the mechanisms involved in thrombotic events in the population with lung cancer, with clear therapeutic impacts.

This is a case-control study with groups differentiated by the presence or absence of NSCLC and matched by age, sex and presence or absence of smoking in the 6 months prior to inclusion. Patients diagnosed with NSCLC without prior treatment for the disease will be candidates for participation in the study.

The primary objective is to compare platelet aggregability by optical aggregometry assessed by the AggRAM® method in patients diagnosed with NSCLC, prior to any oncological treatment, in relation to a control group matched by sex, age and presence or absence of smoking in the previous 6 months. to inclusion Secondary objetives includes laboratorial test of inflammation, coagulation and subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old;
* Confirmed diagnosis of non-small cell lung carcinoma in the case group; absence of history of any neoplasia for control group
* Agreement to sign the Free and Informed Consent Form

Exclusion Criteria:

* Anticoagulation in the last 30 days;
* Use of any antiplatelet agent in the last 30 days;
* Use of any non-steroidal anti-inflammatory drugs in the last 30 days;
* Known platelet dysfunction or platelets <100,000/mm3 or >450,000/mm3;
* Creatinine clearance by MDRD <30 ml/min/1.73 m2
* Eastern Cooperative Oncology Group Performance Status Scale (ECOG) >2
* Known coagulation disorder;
* Hematocrit less than 34% or greater than 55%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Platelet Aggregation analyzed by optical aggregometry-ADP (AggRAM™- Helena Laboratories) | 14 days
  Compare platelet aggregation analyzed by optical aggregometry-ADP (AggRAM™- Helena Laboratórios) between both groups

SECONDARY OUTCOMES:
Platelet aggregability by AggRAM™ ADP after 14 days of use of Clopidogrel 75 mg/day | 14 days
  Evaluation of Platelet aggregability by AggRAM™ ADP after 14 days of use of Clopidogrel 75 mg/day
Platelet aggregability by Plateletworks-ADP at baseline and after 14 days of use of Clopidogrel 75 mg/day | 14 days
  Evaluation of Platelet aggregability by Plateletworks-ADP at baseline and after 14 days of use of Clopidogrel 75 mg/day
Serum levels of tissue factor | Baseline
  Evaluation of Serum levels of tissue factor
Serum levels of type I plasminogen activator inhibitor (PAI 1) | Baseline
  Evaluation of Serum levels of type I plasminogen activator inhibitor (PAI 1)
Serum levels of immature platelets | Baseline
  Evaluation of Serum levels of immature platelets
Serum levels of ultrasensitive C-reactive protein (hs-CRP); | Baseline
  Avaliation of Serum levels of ultrasensitive C-reactive protein (hs-CRP)
Serum levels of interleukin 6 | Baseline
  Evaluation of Serum levels of interleukin 6
Serum levels of Interleukin 1 | Baseline
  Evaluation of interleukin 1
Serum levels of P-Selectin | Baseline
  Evaluation of Serum levels of P-Selectin
Serum levels of D-dimero | Baseline
  Evaluation of Serum levels of D-dimero
Serum levels of Lipoprotein(a) (LPa) | Baseline
  Evaluation of Serum levels of Lipoprotein(a) (LPa)
Serum levels of Glycated hemoglobin | Baseline
  Evaluation of Serum levels of Glycated hemoglobin
Serum levels of coagulogram | Baseline
  Evaluation of Serum levels of coagulogram
Serum levels of Fibrinogen | Baseline
  Evaluation of Serum levels of Fibrinogen
Serum levels of cholesterol ester transfer proteins | Baseline
  Evaluation of Serum levels of cholesterol ester transfer proteins
Serum levels of blood count with platelets | Baseline
  Evaluation of Serum levels of blood count with platelets

OTHER OUTCOMES:
Subgroup Analysis- Age | Baseline and 14 days
  Age (≥65 years or < 65 years)
Subgroup Analysis- Sex | Baseline and 14 days
  Sex (male/female)
Subgroup Analysis- Diabetes mellitus | Baseline and 14 days
  Diabetes mellitus (presence or not)
Subgroup Analysis-Glomerular filtration rate | Baseline and 14 days
  Glomerular filtration rate (CKD EPI) (< 60ml/min/m2 or ≥ 60 ml/min/m2)
Subgroup Analysis- BDI | Baseline and 14 days
  Body Mass Index (<30 or ≥ 30 kg/m2)
Subgroup Analysis- Smoking | Baseline and 14 days
  Current smoking (yes or no)

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor) / University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Fuentes HE, Oramas DM, Paz LH, Casanegra AI, Mansfield AS, Tafur AJ. Meta-analysis on anticoagulation and prevention of thrombosis and mortality among patients with lung cancer. Thromb Res. 2017 Jun;154:28-34. doi: 10.1016/j.thromres.2017.03.024. Epub 2017 Apr 1. PMID 28402864
- [Background] Mutlu H, Artis TA, Erden A, Akca Z. Alteration in mean platelet volume and platicrit values in patients with cancer that developed thrombosis. Clin Appl Thromb Hemost. 2013 Jun;19(3):331-3. doi: 10.1177/1076029611433644. Epub 2012 Feb 16. PMID 22345488
- [Background] Zacharski LR, Henderson WG, Rickles FR, Forman WB, Cornell CJ Jr, Forcier RJ, Edwards RL, Headley E, Kim SH, O'Donnell JF, et al. Effect of warfarin anticoagulation on survival in carcinoma of the lung, colon, head and neck, and prostate. Final report of VA Cooperative Study #75. Cancer. 1984 May 15;53(10):2046-52. doi: 10.1002/1097-0142(19840515)53:103.0.co;2-f. PMID 6322957
- [Background] Ek L, Gezelius E, Bergman B, Bendahl PO, Anderson H, Sundberg J, Wallberg M, Falkmer U, Verma S, Belting M; Swedish Lung Cancer Study Group (SLUSG). Randomized phase III trial of low-molecular-weight heparin enoxaparin in addition to standard treatment in small-cell lung cancer: the RASTEN trial. Ann Oncol. 2018 Feb 1;29(2):398-404. doi: 10.1093/annonc/mdx716. PMID 29106448
- [Background] Macbeth F, Noble S, Evans J, Ahmed S, Cohen D, Hood K, Knoyle D, Linnane S, Longo M, Moore B, Woll PJ, Appel W, Dickson J, Ferry D, Brammer C, Griffiths G. Randomized Phase III Trial of Standard Therapy Plus Low Molecular Weight Heparin in Patients With Lung Cancer: FRAGMATIC Trial. J Clin Oncol. 2016 Feb 10;34(5):488-94. doi: 10.1200/JCO.2015.64.0268. Epub 2015 Dec 23. PMID 26700124
- [Background] Altinbas M, Coskun HS, Er O, Ozkan M, Eser B, Unal A, Cetin M, Soyuer S. A randomized clinical trial of combination chemotherapy with and without low-molecular-weight heparin in small cell lung cancer. J Thromb Haemost. 2004 Aug;2(8):1266-71. doi: 10.1111/j.1538-7836.2004.00871.x. PMID 15304029
- [Background] Meikle CK, Meisler AJ, Bird CM, Jeffries JA, Azeem N, Garg P, Crawford EL, Kelly CA, Gao TZ, Wuescher LM, Willey JC, Worth RG. Platelet-T cell aggregates in lung cancer patients: Implications for thrombosis. PLoS One. 2020 Aug 10;15(8):e0236966. doi: 10.1371/journal.pone.0236966. eCollection 2020. PMID 32776968
- [Background] Navi BB, Reiner AS, Kamel H, Iadecola C, Okin PM, Elkind MSV, Panageas KS, DeAngelis LM. Risk of Arterial Thromboembolism in Patients With Cancer. J Am Coll Cardiol. 2017 Aug 22;70(8):926-938. doi: 10.1016/j.jacc.2017.06.047. PMID 28818202
- [Background] Mangalpally KK, Siqueiros-Garcia A, Vaduganathan M, Dong JF, Kleiman NS, Guthikonda S. Platelet activation patterns in platelet size sub-populations: differential responses to aspirin in vitro. J Thromb Thrombolysis. 2010 Oct;30(3):251-62. doi: 10.1007/s11239-010-0489-x. PMID 20502945
- [Background] Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med. 2000 Mar 27;160(6):809-15. doi: 10.1001/archinte.160.6.809. PMID 10737280
- [Background] Blom JW, Doggen CJ, Osanto S, Rosendaal FR. Malignancies, prothrombotic mutations, and the risk of venous thrombosis. JAMA. 2005 Feb 9;293(6):715-22. doi: 10.1001/jama.293.6.715. PMID 15701913
- [Background] Metharom P, Falasca M, Berndt MC. The History of Armand Trousseau and Cancer-Associated Thrombosis. Cancers (Basel). 2019 Jan 31;11(2):158. doi: 10.3390/cancers11020158. PMID 30708967
- [Background] Marks MA, Engels EA. Venous thromboembolism and cancer risk among elderly adults in the United States. Cancer Epidemiol Biomarkers Prev. 2014 May;23(5):774-83. doi: 10.1158/1055-9965.EPI-13-1138. Epub 2014 Mar 8. PMID 24608188